CLINICAL TRIAL: NCT01200303
Title: Prospective Evaluation of Computer-Assisted, Non-Cathartic CT Colonography for Detection of Adenomatous Colonic Polyps in a Screening Cohort
Brief Title: Evaluation of Computer-assisted, Non-cathartic CT Colonography
Acronym: ncCTC
Status: Completed | Phase: Phase 2 / Phase 3 | Type: Interventional
Sponsor: Massachusetts General Hospital (Other)
Collaborators: GE Healthcare (Industry); American Cancer Society, Inc. (Other)
Responsible Party: Principal Investigator, Michael Zalis MD, Principal Investigator, Massachusetts General Hospital
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Diagnostic
Other Study IDs: GEH-03-OPQ-001; ACS 116256-RSG-08-221-01-CCE (Other Grant/Funding Number: American Cancer Society)
Record Dates: First submitted 2010-09-09; First posted 2010-09-13 (Estimated); Last update posted 2015-08-05 (Estimated); Status verified 2015-08

CONDITIONS: Colonic Polyps
Keywords: colon cancer; adenomatous colonic polyps; colon screening; CT Colonography (Virtual Colonoscopy); Computer Aided Detection; Electronic Cleansing
MeSH Terms: conditions — Colonic Polyps; Colonic Neoplasms | interventions — Iohexol

STUDY DESIGN:
Oversight: Data Monitoring Committee: No

ARMS (1):
- non-cathartic CTC and OC (Active Comparator): This is a single arm, open label, prospective test comparison of non-cathartic, CAD-assisted CTC to segmentally unblinded optical colonoscopy (OC). All study subjects receive both tests, starting with CTC, followed by OC within 5 weeks. CTC results are recorded and revealed to endoscopist on a segment-by-segment basis after initial (blinded) OC evaluation; endoscopist can double check / confirm lesion presence after unblinding and this second read serves as reference standard.
  Interventions: Procedure: non-cathartic CTC

INTERVENTIONS:
Procedure: non-cathartic CTC — non-cathartic, CAD-assisted CT Colonography
  Other Names: tagging of non-cathartic CTC employs iohexol (Omnipaque 300)

SUMMARY:
The purpose of this study is to evaluate the performance of a non-cathartic, computer-assisted form of CT Colonography (Virtual Colonoscopy) for detection of pre-cancerous colon polyps in a group of asymptomatic screening patients.

DETAILED DESCRIPTION:
Examinations to completely assess the colonic anatomy for the purposes of polyp detection and cancer prevention all require an unpleasant, pre-exam cathartic bowel preparation. The discomfort and embarrassment associated with this bowel prep has been identified as a barrier to adherence of at-risk subjects with recommended colon screening guidelines. CT Colonography (CTC) is an imaging based test that evaluates the entire colon anatomy and requires cathartic bowel prep; its performance is considered comparable to optical colonoscopy (OC) for adenomatous polyp detection. In addition, CTC generates a large amount of data to be read by a human, and this data interpretation task can be aided by computer-assisted-detection (CAD) software to identify potential polyp lesions for the human reviewer. This trial studies the performance of a form of CTC that uses fecal tagging and electronic image cleansing to obviate the need for cathartic prep. In addition, readings prospectively employ CAD to potentially buffer human interpretation performance. The investigators are prospectively testing this augmented (non-cathartic, CAD-assisted) form of CTC in asymptomatic (screening) cohort. The trial is a prospective test comparison, using segmentally unblinded optical colonoscopy in combination with pathology specimens as a reference standard for presence of target lesions, adenomatous polyps 6 mm or greater in size.

ELIGIBILITY:
Inclusion Criteria:

* age 50-80, eligible for colon screening

Exclusion Criteria:

* prior anatomic colon screening exam (optical colonoscopy, sigmoidoscopy, barium enema, CT Colonography) within last 5 years
* personal history of inflammatory bowel disease, polyposis syndrome, colo-rectal cancer, colon surgery
* documented passage of blood per rectum within last 12 months

Ages: 50 Years to 80 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Enrollment: 605 (Actual)
Dates: Start 2005-06; Primary Completion 2010-10 (Actual); Study Completion 2011-01 (Actual)

PRIMARY OUTCOMES:
Performance for detection of adenomatous colonic polyps > 6mm | on per subject basis, metric will be assessed at unblinding OC (w/i 5 weeks enrollment); for cohort, summary statistics will be generated at study completion
  this is a prospective test comparison of non-cathartic, CAD-assisted CT Colonography to segmentally unblinded optical colonoscopy (OC), latter serving with pathology specimens as reference standard for presence of polyps.

SECONDARY OUTCOMES:
Patient comfort associated with non-cathartic exam preparation | on per subject basis, outcome will be assessed at 5 weeks post enrollment (following OC); for cohort, summary statistics will be generated at study completion
  as part of the prospective test comparison, we are generating summary statistics of self-reported patient comfort assessments with the test (non-cathartic) exam preparation versus standard, cathartic preparation.

CONTACTS AND LOCATIONS:
Overall Officials: Michael Zalis, MD, Principal Investigator — Massachusetts General Hospital
Locations (3):
- United States (3):
  - UCSF-VA Medical Center, San Francisco, California
  - Massachusetts General Hospital, Boston, Massachusetts
  - Brigham and Women's Hospital, Boston, Massachusetts

REFERENCES:
- [Result] Zalis ME, Blake MA, Cai W, Hahn PF, Halpern EF, Kazam IG, Keroack M, Magee C, Nappi JJ, Perez-Johnston R, Saltzman JR, Vij A, Yee J, Yoshida H. Diagnostic accuracy of laxative-free computed tomographic colonography for detection of adenomatous polyps in asymptomatic adults: a prospective evaluation. Ann Intern Med. 2012 May 15;156(10):692-702. doi: 10.7326/0003-4819-156-10-201205150-00005. PMID 22586008